CLINICAL TRIAL: NCT05582460
Title: Exploring the Value of the Reporter Gene Assay and Flow Cytometry of Synovial Fluid in Total Hip and Knee Arthroplasty as a Diagnostic Tool for Periprosthetic Joint Infection
Brief Title: Exploring Novel Diagnostic Tools for Periprosthetic Joint Infection
Acronym: VECTOR-PJI
Status: Completed | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-2054
Record Dates: First submitted 2022-10-13; First posted 2022-10-17 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Prosthesis-Related Infections; Arthroplasty, Replacement, Hip; Arthroplasty, Replacement, Knee
MeSH Terms: conditions — Prosthesis-Related Infections | interventions — Flow Cytometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PJI: Patients diagnosed with a PJI based on the EBJIS criteria ('Infection confirmed')
  Interventions: Diagnostic Test: Reporter Gene Assay; Diagnostic Test: Flow Cytometry
- No PJI: Patients not diagnosed with a PJI based on EBJIS criteria
  Interventions: Diagnostic Test: Reporter Gene Assay; Diagnostic Test: Flow Cytometry

INTERVENTIONS:
Diagnostic Test: Reporter Gene Assay — Transcription factor reporter gene assay using luciferase
Diagnostic Test: Flow Cytometry — Flow Cytometry Analysis using the Sysmex UF-4000, analyzing for bacteria, mononuclear and polymorphonuclear cells, and red blood cell and white blood cell count.

SUMMARY:
Joint replacement is a valuable surgical intervention that improves quality of life, provides pain relief, and restores function of patients. However, some patients need revision surgery due to failure of the implant, with periprosthetic joint infection (PJI) remaining a rare but serious complication following total hip (THA) and knee (TKA) arthroplasty. Diagnosing PJI is a major challenge as no diagnostic test with absolute accuracy exists. The diagnosis is based on a combination of clinical findings, laboratory results from peripheral blood and synovial fluid, microbiological culture, histological evaluation of periprosthetic tissue, and intraoperative findings. However, the preoperative diagnosis can be inconclusive and operative criteria are required for the definitive diagnosis. Therefore, novel diagnosing tools for identification of PJI are necessary.

A recent study using a gene reporter assay, identified biomarkers in synovial fluid that define joint states in patients with osteoarthritis.However, no previous studies have investigated cellular signaling in synovial fluid of patients with PJI. With this study we want to explore the potential of a reporter gene assay of synovial fluid in patients with PJI and without PJI of their TKA and THA.

Also, flow cytometry analysis of biological fluids has recently received increased attention as a potentially valuable method in diagnosing infections. For example, the method is already used to analyze urine samples for urinary tract infections. Recently, researchers have now also used this method to screen for the presence of bacteria. The most important limitation of flow cytometry analysis of synovial fluids for bacteria to date is that it is unclear as to which bacteria count value - the cutoff value - represent patients with PJI and which represent patients without PJI. With this study we want to explore the potential of flow cytometry analysis of synovial fluid in categorizing patients with PJI and without PJI.

Our primary objective is to explore the value of synovial fluid analysis using a reporter gene assay and flow cytometry in the detection of a periprosthetic joint infection.

ELIGIBILITY:
Inclusion Criteria:

* All patients planned for elective THA or TKA revision surgery with revision of one or more fixed components will be eligible to participate in this study.

Exclusion Criteria:

* are planned for a revision of single mobile parts only;
* have received intravenous and/or oral antibiotics within 2 weeks before the diagnostic workup and/or surgery;
* are unable to provide their consent for use of their human tissues for medical research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients visiting the outpatient clinic of the participating hospitals and planned for elective revision surgery of their THA or TKA.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2025-07-23 (Actual)

PRIMARY OUTCOMES:
Fold change of luciferase assay | Within 30 days of surgery
  Diagnostic performance of the reporter gene assay of synovial fluid by calculating fold change data from the reporter gene measurements.
  A luciferase assay will be performed using the collected synovial fluid and the amount of luciferase activity will be measured by luminometer and expressed in relative light units (RLU). A background control (e.g., medium or buffer alone) will be used to evaluate raw RLU values that will be subtracted from all the sample values for better accuracy. The data for the reporter assay will be expressed using an equation to determine normalized fold change in activity between the two groups.
Diagnostic performance of flow cytometric analysis | Within 4 hours of surgery
  Diagnostic performance of the flow cytometry analysis of synovial fluid by determining difference in results between two groups using ROC curve analysis.
  If a cut-off point has been determined, sensitivity (SN), specificity (SP), negative (NPV) and positive predictive value (PPV) can be calculated.

SECONDARY OUTCOMES:
Sensitivity of the flow cytometric analysis | Within 4 hours of surgery
Specificity of the flow cytometric analysis | Within 4 hours of surgery
Positive predictive value of the flow cytometric analysis | Within 4 hours of surgery
Negative predictive value of the flow cytometric analysis | Within 4 hours of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Rijnstate Hospital, Arnhem, Gelderland, Netherlands